CLINICAL TRIAL: NCT00324883
Title: Urine Chloride/Creatinine Ratio for Estimation of Urine Sodium
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Allied Minds (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0601008328
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Hypertension
Keywords: sodium intake; sodium excretion; chloride excretion; creatinine; hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No

SUMMARY:
We plan to assess the accuracy of a new means of estimating urine sodium excretion. We will compare the chloride to creatinine ratio obtained by titrator sticks with urine sodium measured by a standard laboratory. If found to approximate sodium excretion, the titrator sticks could provide a convenient means for doctors and patients to monitor their salt intake.

DETAILED DESCRIPTION:
Level of salt intake has an important impact in patients with high blood pressure or congestive heart failure. Despite this there is no convenient way for doctors or patients to assess their salt intake other than diet recall, which is unreliable, or measurement of sodium excretion in a 24 hour collection of urine, which is very inconvenient. As a result, salt intake is not monitored in most patients.

2 innovations might enable a more convenient assessment of salt intake. A titrator stick that measures chloride ion concentration (chloride and sodium concentrations correlate strongly with each other), and a titrator stick that measures urine creatinine. The latter enables estimation of 24 hour excretion from a single sample of urine. In assessing sodium intake, a measurement that provides an approximation of urine sodium intake would be of considerable clinical value

In this study, we shall compare the estimation of urine sodium excretion measured by a laboratory with estimation of sodium excretion from measurement of chloride/creatinine ration in a random urine sample. We will compare the estimate obtained by titrator stick with the sodium concentration from the same urine sample, and from measurements obtained from a 24 hour urine collection. In the next phase we will also compare the average estimate from titrator stick obtained on 3 different days with the measurement obtained from 3 24 hour urine collections.

We will assess the accuracy with which the titrator stick estimate approximates the measured urine sodium.

As of March 2007, we have recruited 50 subjects, and continue to study the predictive value of spot urine chloride/creatinine ratio, as described.

ELIGIBILITY:
Inclusion Criteria:

Over 21 years of age.

Exclusion Criteria:

No exclusion criteria.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: volunteers from patient population including hypertensive and normotensive individuals, and hypertensive and normotensive volunteers recruited by advertising. Age >21 excluding individuals with unstable changes in renal function.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2006-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
urine sodium excretion | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Samuel J Mann, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College of Cornell University, New York, New York, United States